CLINICAL TRIAL: NCT04772352
Title: Effects of Febuxostat for Interventions of Lowering Uric Acid in Patients With Gout With Nonalcoholic Fatty Liver Disease: a Multicenter, Open-label, Randomized, Controlled Study
Brief Title: Effects of Febuxostat for Lowering Uric Acid in NAFLD Patients With Gout
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUANAFLD V1.0
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: A total of 200 subjects are enrolled in this study. After the initial screening, the subjects were randomly divided into the control group and the drug treatment group. The control group was given lifestyle intervention at 0-24 weeks, and the experimental group was given febuxostat oral therapy on the basis of lifestyle intervention. If the results showed that the reduction of liver fat content of subjects in the lifestyle intervention combined with febuxostat treatment group was significantly better than that in the lifestyle intervention group alone, the original intervention was continued in the drug treatment group, and the control group was given febuxostat orally on the basis of the lifestyle intervention at 24-48 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Lifestyle intervention + febuxostat (40mg, once a day, orally) (Experimental): participants accept febuxostat treatment in addition to lifestyle intervention for 0-48 week.
  Interventions: Drug: febuxostat treatment; Behavioral: lifestyle intervention
- Control group: Lifestyle intervention (Active Comparator): participants receive lifestyle intervention for 0-24 week. If the results of the 0-24 week study showed that the liver fat content of subjects in the experimental group was significantly lower than that in the control group, control group will accept febuxostat treatment in addition to lifestyle intervention in the next 25-48 week.
  Interventions: Behavioral: lifestyle intervention

INTERVENTIONS:
Drug: febuxostat treatment — According to NAFLD guidelines, participants accept febuxostat treatment (40mg, once a day, orally)
  Arms: Experimental group: Lifestyle intervention + febuxostat (40mg, once a day, orally)
Behavioral: lifestyle intervention — According to NAFLD guidelines, participants receive lifestyle intervention (diet and exercise).

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common and harmful chronic liver disease. NAFLD accounts for 49.3% of the total number of chronic liver disease patients in China. It is important to effectively prevent and control NAFLD and its related diseases.

Previous studies show the level of serum uric acid is significantly elevated in patients with NAFLD. Xanthine oxidase is a key enzyme in uric acid metabolism. It is a new therapeutic target for NAFLD.

This study is aimed to further confirm that hyperuricemia is a new risk factor for NAFLD through a large sample prospective study. Furthermore, this study explore whether Xanthine oxidase (XO), a key enzyme in uric acid metabolism, plays an important role in regulating NAFLD.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common and harmful chronic liver disease. NAFLD accounts for 49.3% of the total number of chronic liver disease patients in China. It is important to effectively prevent and control NAFLD and its related diseases.

Previous studies show the level of serum uric acid is significantly elevated in patients with NAFLD. In a large cross-sectional study, the researcher were the first to confirm that serum uric acid level was significantly increased in patients with NAFLD. The results were published in J Hepatol. Xanthine oxidase is a key enzyme in uric acid metabolism. It is a new therapeutic target for NAFLD.

This study is aimed to further confirm that hyperuricemia is a new risk factor for NAFLD through a large sample prospective study. Furthermore, this study explore whether Xanthine oxidase (XO), a key enzyme in uric acid metabolism, plays an important role in regulating NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* with informed consent;
* Ages 18-65;
* Overweight/obesity: BMI ≥24kg/m2;
* A history of gout with serum uric acid levels of > 420μmol/L in men and postmenopausal women, and >360 μmol/L in premenopausal women;
* Moderate or above fatty liver was found in the initial screening by ultrasound, and the liver fat content was more than 15% as determined by MRI-PDFF.

Exclusion Criteria:

* with a history of allergy to febuxostat and allopurinol;
* in the acute active phase of gout;
* Drinking equivalent to alcohol intake ≥30g/d(male), ≥20g/d(female);
* Patients with obvious abnormal liver function: serum transaminase (ALT, AST, GGT one of them) or serum bilirubin (direct bilirubin, indirect bilirubin one of them) exceed 2 times the upper limit of normal reference value; Serum albumin <35g/L;
* Have a history of viral hepatitis, or serological examination suggests hepatitis virus infection, or have a history of other liver diseases;
* Complicated with renal insufficiency (SCr >133μmol/L) or urinary protein +;
* Complicated coronary heart disease;
* Cardiac dysfunction (cardiac function grade 2 or above);
* Complementation with diabetes, or fasting blood glucose >7.8mmol/L, or HbA1c >7.5%;
* Severe hypertension, blood pressure ≥ 160/100 mmHg;
* Patients with asthma and other respiratory diseases;
* Intestinal diseases such as inflammatory bowel disease;
* Any history of systemic malignancy in the past 5 years;
* Morbid obesity (BMI>37.5kg/m2);
* Triglyceride ≥5.0 mmol/L was found to be significantly abnormal in baseline examination;
* had received systemic hormone or immunosuppressive therapy within 3 months prior to screening, or expected to receive hormone or immunosuppressive therapy in the future;
* Use of uric-lowering drugs in the 4 weeks before screening: febuxostat, benzobromarone, allopurinol;
* Use of other drugs affecting uric acid metabolism were adjusted within 4 weeks before screening: losartan, fenofibrate, irbesartan, thiazide diuretics, loop medullaral diuretics, compound antihypertensive agents containing diuretics;
* Other drugs that may affect liver fat content were taken within 4 weeks before screening;
* Weight change ≥5% within 3 months before screening;
* Women who are lactating or pregnant or who plan to become pregnant within one year;
* were enrolled in other studies within 6 months before screening;
* unsuitable for participants to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Liver fat content of subjects in different groups | at the first week.
  Liver fat was assessed based on Magnetic Resonance Imaging (MRI).
Liver fat content of subjects in different groups | at the 24th week .
  Liver fat was assessed based on Magnetic Resonance Imaging (MRI).
Liver fat content of subjects in different groups | at the 48th week.
  Liver fat was assessed based on Magnetic Resonance Imaging (MRI).
Serum uric acid levels of subjects in different groups | at the first week
  blood samples was assessed after 12 hours overnight fasting for the determination of hematological and biochemical variables, which were measured using an automated hematology analyzer by standard methods.
Serum uric acid levels of subjects in different groups | at the forth week.
  blood samples was assessed after 12 hours overnight fasting for the determination of hematological and biochemical variables, which were measured using an automated hematology analyzer by standard methods.
Serum uric acid levels of subjects in different groups | at the twelfth week.
  blood samples was assessed after 12 hours overnight fasting for the determination of hematological and biochemical variables, which were measured using an automated hematology analyzer by standard methods.
Serum uric acid levels of subjects in different groups | at the 24th week.
  blood samples was assessed after 12 hours overnight fasting for the determination of hematological and biochemical variables, which were measured using an automated hematology analyzer by standard methods.
Serum uric acid levels of subjects in different groups | at the 36th week.
  blood samples was assessed after 12 hours overnight fasting for the determination of hematological and biochemical variables, which were measured using an automated hematology analyzer by standard methods.
Serum uric acid levels of subjects in different groups | at the 48th week.
  blood samples was assessed after 12 hours overnight fasting for the determination of hematological and biochemical variables, which were measured using an automated hematology analyzer by standard methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No